CLINICAL TRIAL: NCT02259933
Title: A Double-blind (at Each Dose Level), Randomised, Placebo Controlled Study to Evaluate Safety, Tolerability and Pharmacokinetics of Increasing Repeated Oral Doses of KUC 7483 CL Tablets (Dosage: 40, 120, 180 mg b.i.d.) Over 7 Days in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of KUC 7483 CL Tablets in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1207.3
Record Dates: First submitted 2014-10-07; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- KUC 7483 CL (Experimental): increasing repeated oral doses
  Interventions: Drug: KUC 7483 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KUC 7483 CL
  Arms: KUC 7483 CL
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability and pharmacokinetics of KUC 7483 CL after repeated dosing

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
   * No finding deviating from normal and of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥21 and Age ≤60 years
3. BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
3. History of relevant orthostatic hypotension, fainting spells or blackouts
4. Chronic or relevant acute infections
5. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
6. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
7. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
8. Participation in another trial with an investigational drug within two months prior to administration or during the trial
9. Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
10. Inability to refrain from smoking on trial days
11. Alcohol abuse (more than 60 g/day)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range of clinical relevance

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2004-02; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal findings in physical examination | up to 8 days after last drug administration
Number of subjects with clinically significant changes in 12-lead ECG (electrocardiogram) | up to 8 days after last drug administration
Number of subjects with clinically significant changes in vital signs | up to 8 days after last drug administration
  Blood Pressure, Pulse Rate, body temperature, orthostatic testing
Number of subjects with clinically significant changes in laboratory tests | up to 8 days after last drug administration
Changes in salivary secretion | pre-dose and 2, 4 and 8 hours after drug administration on days 1 and 7
Changes in residual urine volume | pre-dose and 2, 4 and 8 hours after drug administration on days 1 and 7
Number of subjects with adverse events | up to 8 days after last drug administration
Assessment of tolerability by investigator on a 5-point scale | within 8 days after last drug administration
Number of subjects with clinically significant changes in special laboratory parameters | up to day 8
  Tropanin I, Insulin, C-Peptide, Glucagon, free fatty acids and faecal occult blood testing, Potassium, Lactate and cAMP

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | up to day 9
Time from dosing to the maximum concentration of the analyte in plasma (Tmax) | up to day 9
Area under the concentration-time curve of the analyte in plasma (AUC) | up to day 9
Terminal rate constant of the analyte constant in plasma (λz) | up to day 9
Terminal half-life of the analyte in plasma (t1/2) | up to day 9
Mean residence time of the analyte in the body after oral administration (MRTpo) | up to day 9
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | up to day 9
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | up to day 9
Amount of the analyte that is eliminated in urine from the time point t1 until time point t2 (Aet1-t2) | up to day 9
Fraction of administered drug excreted in urine from the time point t1 until time point t2 (fet1-t2) | up to day 9
Renal clearance of the analyte determined from the time point t1 until time point t2 (CLR,t1-t2) | up to day 9
Minimum concentration of the analyte in plasma at steady state (Cmin,ss ) | up to day 9
Accumulation ratio (RA) | up to day 9
Linearity index (LI) | up to day 9